CLINICAL TRIAL: NCT03325296
Title: Efficacy of Twice Daily Application of LEO 124249 Ointment 30 mg/g for 12 Weeks on Eyebrow Alopecia Areata.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXP-1377; 2017-002720-24 (EudraCT Number)
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2018-07

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Ointments

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LEO 124249 ointment 30 mg/g (Experimental): Ointment to be applied on the eyebrow twice daily.
  Interventions: Drug: LEO 124249
- LEO 124249 ointment vehicle (Placebo Comparator): Ointment to be applied on the eyebrow twice daily.
  Interventions: Other: Ointment vehicle

INTERVENTIONS:
Drug: LEO 124249 — Ointment containing LEO 124249
  Arms: LEO 124249 ointment 30 mg/g
Other: Ointment vehicle — Ointment without active ingredients
  Arms: LEO 124249 ointment vehicle

SUMMARY:
This clinical trial attempts to investigate the efficacy of LEO 124249 ointment in the treatment of alopecia areata on the eyebrows.

ELIGIBILITY:
Inclusion Criteria:

* Clinical unequivocal diagnosis of Alopecia Areata (patchy, univeralis and totalis), on both scalp and eyebrows as assessed by the investigator.
* Maximal disease duration of current episode of Alopecia Areata on the eyebrows of 3 years at screening.
* Maximal Alopecia Areata disease duration - defined as years of active disease - in other locations than eyebrows of 10 years at screening.

Exclusion Criteria:

* Clinical diagnosis of diffuse type alopecia areata as assessed by the investigator.
* Any topical, intralesional therapy or procedure applied within 2 cm of the treatment area, within 4 weeks of randomisation, which in the opinion of the investigator, could interfere with the trial assessments. This includes, but is not limited to: corticosteroids, calcineurin inhibitors, calcipotriol, minoxidil, antimicrobials, prostaglandin analogs (e.g. bimatoprost), herbal extracts, topical immunotherapy with allergens or irritants and any laser or phototherapy, and eyebrow tattoo.
* Any systemic treatment with immunosuppressive drugs (e.g. methotrexate, cyclosporine, azathioprine), chloroquin derivatives, corticosteroids (including intralesional treatment outside the trial treatment area), or any other systemic therapy that in the opinion of the investigator could affect hair regrowth, within 4 weeks prior to randomisation.
* Any biologic medicinal product targeting the immune system within 5 half-lives and minimum 4 weeks prior to randomisation (e.g. anti-TNFα, anti-IL17, anti IL12/23, anti IL-4Rα targeting drugs).
* Systemic JAK inhibitor Ruxolitinib (Jakafi®/Jakavi®), Tofacitinib (Xeljanz®) at any time prior to randomisation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 12 of investigator evaluated overall area score (ASoverall L+R) of eyebrow hair growth. | baseline to week 12
  The percentage area of the identified left and right eyebrow area and left and right region of interest (ROI) covered by hair growth will be scored according to the following:
  1-10 % - 1 11-20 % - 2 21-30 % - 3 31-40 % - 4 41-50 % - 5 51-60 % - 6 61-70 % - 7 71-80 % - 8 81-90 % - 9 91-100 % - 10

SECONDARY OUTCOMES:
Treatment emergent AEs (including AEs relating to local tolerability) | baseline to week 12
Degree of response in change from baseline to Week 12 for ASoverall L+R | baseline to Week 12
  Complete response - ≥ 8 Partial response - 4-<8 Minimal response - 1-<4 No response - <1
Investigator evaluation of cosmetic outcome at Week 12 as assessed by Cosmetic outcome Score | baseline to Week 12
  Is the appearance of the eyebrows cosmetically normal and acceptable? Yes - 1 No - due to insufficient regrowth area - 2 No - due to insufficient density - 3 No - due to uneven distribution - 4 No - due to other reason (explain, including combination of the above) - 5

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — LEO Pharma
Locations (2):
- Denmark (2):
  - Investigational site, Aarhus
  - Investigational site, Gentofte Municipality

IPD SHARING:
Plan to Share IPD: No